CLINICAL TRIAL: NCT00823355
Title: A Phase I, Open Label, Dose Ascending Study of BCX1777 (Oral) in Patients With Recurrent or Refractory T/NK-cell Malignancies
Brief Title: Oral Forodesine Hydrochloride (BCX-1777) in Patients With Recurrent or Refractory T/NK-cell Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mundipharma K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BCX1777-J01
Record Dates: First submitted 2009-01-08; First posted 2009-01-15 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Recurrent or Refractory T/NK-cell Malignancies
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BCX1777 (Experimental)
  Interventions: Drug: forodesine hydrochloride

INTERVENTIONS:
Drug: forodesine hydrochloride — Cohort 1: 100mg / body (1 x 100mg tablet once daily)
Drug: forodesine hydrochloride — Cohort 2: 200mg / body (2 x 100mg tablets once daily)
Drug: forodesine hydrochloride — Cohort 3: 300mg / body (3 x 100mg tablets once daily)
Drug: forodesine hydrochloride — Cohort 4: 400mg / body (4 x 100mg tablets once daily)

SUMMARY:
Primary objectives are to evaluate the safety profile and tolerability of oral BCX1777 in each cohort of patients with recurrent or refractory T/NK-cell malignancies and to evaluate pharmacokinetics (PK) of oral BCX1777.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented with histopathological diagnosis from biopsy, T/NK-cell malignancies (WHO classification). Precursor T-cell lymphoblastic leukemia/lymphoma (T-ALL/T-LBL) should be excluded in this study
* A patient with recurrent, relapse or refractory T/NK-cell malignancies who has received at lease one chemotherapeutic regimen
* Age 20 or greater
* Eastern Cooperative Oncology Group(ECOG) performance status:0,1.
* Able to be hospitalized at least for 15 days from the first dose
* In the case of subject with tumor cell rate of ≤25% in bone marrow, a patient who satisfies both of the following criteria.

  * Neutrophil count: ≥1,200/mm3
  * Platelet count: ≥75,000/mm3

    * In the case of CTCL, the tumor cell rate is handled as ≤25%.
* Adequate Liver function: AST, ALT ≤ 5.0 x upper limit of normal (ULN)
* Adequate Renal function: Creatinine Clearance (using cockcroft-Gault formula) ≥ 50mL/min
* Life expectancy of at least 3 months
* A patient who has given a written informed consent prior to the start of procedures proper to this study.

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-01; Primary Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety profile and tolerability of oral BCX1777 in patients with recurrent or refractory T/ NK-cell malignancies. | March 2010
To evaluate pharmacokinetics (PK) of oral BCX1777 | March 2010

SECONDARY OUTCOMES:
To evaluate pharmacodynamics (PD) of oral BCX1777 | March 2010
To correlate the plasma level of BCX1777 with plasma 2'-deoxyguanosine (dGuo) | March 2010
To evaluate the efficacy of oral BCX1777 | March 2010
To analyze cell surface marker in peripheral blood mononuclear cell | March 2010

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Investigational Site, Nagoya, Aichi-ken
  - Investigational Site, Nagasaki, Nagasaki
  - Investigational Site, Cyuo, Tokyo

REFERENCES:
- [Derived] Ogura M, Tsukasaki K, Nagai H, Uchida T, Oyama T, Suzuki T, Taguchi J, Maruyama D, Hotta T, Tobinai K. Phase I study of BCX1777 (forodesine) in patients with relapsed or refractory peripheral T/natural killer-cell malignancies. Cancer Sci. 2012 Jul;103(7):1290-5. doi: 10.1111/j.1349-7006.2012.02287.x. Epub 2012 Apr 30. PMID 22448814